CLINICAL TRIAL: NCT04893473
Title: New Method for Real-time Detection of Tissue Ischemia; IscAlert™ - Study
Brief Title: New Method for Real-time Detection of Tissue Ischemia
Acronym: ISCALERT
Status: Withdrawn | Type: Observational
Why Stopped: Send in by another researcher. This is terminated to avoid two identical studies
Sponsor: Oslo University Hospital (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Espen Lindholm, Principal investigator, Oslo University Hospital
Other Study IDs: 1-20
Record Dates: First submitted 2020-08-10; First posted 2021-05-19 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Ischemia; Blood Circulation Disorder; Carbon Dioxide; Biosensing Techniques
Keywords: Ischemia; Carbon dioxide; Biosensor; Musculature; Subcutaneous; Surgery; Orthopedic; Limb
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients scheduled for limb (arm/leg) surgery with tourniquet where IscAlert is removed immediately after surgery.
  All patients will receive 3 sensors in the limb undergoing surgery and two control sensors in the opposite limb. The sensor in the opposite extremity which is not to be operated serves as a reference value for carbon dioxide.
  Interventions: Device: IscAlert
- Group 2: Patients scheduled for limb (arm/leg) surgery with tourniquet where IscAlert is removed 72 hours after surgery.
  All patients will receive 3 sensors in the limb undergoing surgery and two control sensors in the opposite limb. The sensor in the opposite extremity which is not to be operated serves as a reference value for carbon dioxide.
  Interventions: Device: IscAlert

INTERVENTIONS:
Device: IscAlert — 3 IscAlert sensors in the limb undergoing surgery and two control sensors in the opposite limb are inserted and carbon dioxide is measured continuously.

SUMMARY:
This is a prospective, single arm, open, single centre clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for limb (arm/leg) surgery with tourniquet. IscAlert is measuring carbon dioxide in muscular and subcutaneous tissue. IscAlert is inserted into normal muscle and subcutaneous tissue in ischemic (operated limb with a tourniquet) and non-ischemic limb (non-operated limb).After the tourniquet is inflated, ischemia develops in the muscles and subcutaneous tissue. This will result in an increase in carbon dioxide, which will be detected by the sensor on the operated extremity, while the sensor on the non-operated will show normal values. After releasing the tourniquet cuff, the muscle will be reperfused and the carbon dioxide level is expected to decrease into normal levels. 50 number of patients will be enrolled to undergo the procedures. The IscAlert will be removed from the patient before the patient is discharged from the operating room, but in 25 of the patients, IscAlert™ will be inserted for 72 hours in the operated extremity after the end of surgery. After this, the sensors are removed.250 Devices is planned to be used in this clinical study.

DETAILED DESCRIPTION:
This is a prospective, single arm, open, single centre clinical investigation designed to examine the feasibility and safety of the IscAlert™ device in patients scheduled for limb (arm/leg) surgery with tourniquet.

50 number of patients will be enrolled to undergo the procedures detailed in this clinical investigational plan using 250 devices.

IscAlert is 0.8 mm in diameter and in vitro testing, shows stable and accurate measurements of tissue carbon dioxide . More than 100 animal experiments have been done with the sensor. The experiments have shown that the sensor detects ischemia (Increased carbon dioxide-measurements) in real time in the following organs and tissues: Brain, heart, liver, kidneys, pancreas, intestines, musculature and subcutaneous tissue. Sensitivity and specificity are close to 100%. The sensors are inserted into tissue by a split needle technique. The split needle is the size of a 3-gauge peripheral venous catheter. In animal studies, no complications have been detected when using the sensor.

The IscAlert catheters are connected to an electronics unit that is fixed to the skin with an adhesive plaster outside the sterile area. The electrical signals are redirected to a personal computer approved for clinical use which continuously records tissue pressures of carbon dioxide .

IscAlert is inserted into normal muscle and subcutaneous tissue proximal on the limb to be operated. The insertion is distal to the blood cuff, and far away from the surgery field. The insertion is done under sterile conditions in accordance with standard sterility criteria at the hospital. No pain during insertion will occur because of insertion is performed after anesthesia induction. Also, the insertion can be compared to an intramuscular injection.

An identical IscAlert catheter is also inserted in the opposite extremity that is not to be operated and serves as a reference value. After the tourniquet is inflated, ischemia develops in the muscles and subcutaneous tissue. This will result in an increase in carbon dioxide, which will be detected by the sensor on the operated extremity, while the sensor on the non-operated will show normal values.

After releasing the tourniquet cuff, the muscle will be reperfused and the carbon dioxide level is expected to decrease into normal levels within 15 - 45 minutes. In 25 patients, the biosensors will be removed from the patient before the patient is discharged from the operating room, but in 25 of the patients, IscAlert will be inserted for 72 hours in the operated extremity after the end of surgery to identify drifting of the sensors. After this, the sensors are removed.

The primary objective is to evaluate the ability of the IscAlert device to measure carbon dioxide levels in ischemic and non-ischemic limb musculature and subcutaneous tissue in patients who experience orthopedic surgery with limb tourniquet and to assess the safety/efficacy using device IscAlert.

Our hypotheses are:

1. The IscAlert device will be able to detect the presence of ischemia in muscle and subcutaneous tissue, whereby carbon dioxide levels, measured by IscAlert, will be higher in ischemic musculature than non-ischemic musculature in patients undergoing orthopedic limb surgery.
2. No clinically significant bleeding or infection will occur using IscAlert in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be scheduled for orthopedic limb surgery with planned use of tourniquet.
* Subject must be ≥ 18 years
* Able to give written signed informed consent
* Tourniquet planned to be used > 30 minutes

Exclusion Criteria:

* Sign of inflammation/infection, hematoma, and traumatized tissue at insertion site
* Chronic use of anticoagulants

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need limb surgery with tourniquet cuff
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-14 (Estimated); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Tissue carbon dioxide level | 72 hours
  Tissue carbon dioxide level (kPa) during insertion period

SECONDARY OUTCOMES:
Bleeding | 72 hours
  Amount of blood from insertion site (ml)
Infection | 1 week
  Infection from insertion site at the discretion of the investigator (yes or no)
Arterial carbon dioxide level | 2 hours
  Blood gass analysis of carbon dioxide during surgery (kPa)
Arterial lactate level | 2 hours
  Blood gass analysis of lactate during surgery (mmol/L)
Arterial pH level | 2 hours
  Blood gass analysis of pH during surgery
Arterial Oxygen level | 2 hours
  Blood gass analysis of Oxygen during surgery (Kpa)
Time of tourniquet | 2 hours
  Minutes of inflated tourniquet during surgery (minutes)
End-tidal level of carbon dioxide | 2 hours
  End-tidal level of carbon dioxide during anesthesia (kPa)

CONTACTS AND LOCATIONS:
Overall Officials: Magne Røkkum, Md, Ph.d, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers